CLINICAL TRIAL: NCT03975322
Title: Prospective Prediction of Malignant Transformation of Oral Leukoplakia Using a MAGE-A-based Immunoscore
Brief Title: Prediction of Malignant Transformation of Oral Leukoplakia Using a MAGE-A-based Immunoscore
Acronym: PREDICT-OLP
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Manuel Weber, Dr. med. Dr. med. dent. Manuel Weber, MD, DMD, Principal Investigator, University of Erlangen-Nürnberg Medical School
Other Study IDs: 1.4
Record Dates: First submitted 2019-05-27; First posted 2019-06-05 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Oral Leukoplakia; Oral Leukoplakia of Tongue; Oral Leukoplakia of Gingiva; Oral Lichen Planus
Keywords: OLP; oral cancer; OSCC; oral squamous cell carcinoma
MeSH Terms: conditions — Leukoplakia, Oral; Lichen Planus, Oral; Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — paraffin specimens and RNAlater specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral squamous cell carcinomas (OSCC) is among the most common malignancies worldwide. Early detection and prevention of OSCC is thought to have the highest potential to reduce morbidity and mortality. In prevention, the main focus is on precancerous lesions, especially oral leukoplakia (OLP), as up to 67% of OSCC arise on the basis of OLP. The determination of the transformation risk of OLP by histological determination of the degree of dysplasia is unreliable.

A promising marker for the timely development of a OSCC is the detection of antigens of the MAGE-A gene family. The special feature of MAGE-A is that they can be detected in 93% of all OSCC and in approx. 85% of OLP that transform to OSCC. The detection of MAGE-A could also indicate changes in the immunological environment that occur prior to malignant OLP transformation and could be used for immunotherapies.

Aim of this study is to investigate MAGE-A as a predictive marker for the malignant transformation of OLP in the setting of a prospective, multicenter study and to establish it as a diagnostic parameter in addition to classical histology. In addition, the association of MAGE-A expression with the occurrence of immunological changes in OLP will be investigated in order to evaluate the possibility of minimally invasive immunotherapy of OLP.

The study is intended to include 500 biopsies of non-selected patients with OLP from university institutions and private practices. The follow-up should be at least 3 years, whereby it is examined whether an OSCC on the basis of the original OLP developed. After three years, an interim evaluation of the results with statistical evaluation will be carried out. In order to ensure that the course of the disease is monitored for at least three years for all OLPs, an extension of the monitoring period to 5 years is planned.

The study could establish a routine diagnostic parameter to supplement the histo-morphological diagnosis of OLP and evaluate the possibility of immunotherapy of OLP.

DETAILED DESCRIPTION:
Oral squamous cell carcinomas (OSCC) is among the most common malignancies worldwide. Despite the introduction of microsurgical reconstruction options and advances in multimodal tumor therapy, the prognosis has not improved significantly in the last 30 years.

The most important aspect for increasing survival rate is seen in the early detection of OSCC and its precursor lesions. Up to 67 % of OSCC develop on the basis of oral leukoplakia (OLP), which frequently occur prior to the diagnosis of carcinoma. OLP treatment depends on the risk of malignant transformation. Therapeutic approaches range from simple observation to complete surgical excision of OLP. The scientific evidence regarding the handling of OLP is low. Current literature outlines missing evidence in therapeutic management of OLP. The early identification of OLP with a high risk of malignant degeneration is a relevant clinical question, since approx. 2% of OLPs transform malignantly each year. In lesions with dysplasia this rate increases to about 17%.

Gold standard for determining the risk of malignant transformation of OLP is the histologic determination of the degree of dysplasia. As the histological degree of dysplasia increases, so does the risk of developing PECM on the basis of OLP. The decision for a surgical or a conservative therapy currently depends on the degree of dysplasia of the OLP. The histopathological assessment of the degree of dysplasia is subjective and depends on the experience of the pathologist making the assessment. However, the major disadvantage in assessing the malignant transformation potential with this method is that many precursor lesions do not follow the histopathologically determined degree of dysplasia. Thus, 0-3% of hyperplasias (D0) and up to 30% of mild dysplasias (D1) transform to OSCC. D0 OLP are lesions, which are usually only observed according to current therapy recommendations. Thus, an assessment of the dignity of OLP and a long-term prediction of the risk for the development of OSCC are not reliable. OLP with a histopathologically low malignancy potential but a cell-biologically probable malignant transformation must be identified in order to prevent undertreatment of these patients.

The aim of this explorative study is to investigate whether the malignant transformation of OLP can be reliably predicted using immunohistochemical and molecular biological methods. A significant association of the expression of MAGE-A expression with the malignant transformation of OLP to OSCC has already been demonstrated in retrospective studies. It is now necessary to further develop these available test procedures and evaluate them in a prospective study in order to transfer them into clinical routine. Sensitivity and specificity of the investigated markers will be investigated in a prospective, multicenter setting. A non-selected group of patients will be examined. The aim is to establish a test procedure that can be used cost-effectively. The MAGE-A expression should serve as an indicator and for the application of new, innovative therapy concepts such as the immunotherapy of OLP.

The following questions will be answered:

i) Do OLP with malignant transformation show an increased MAGE-A expression in a time interval of 3 years (follow-up up to 5 years)? ii) How high is the sensitivity and specificity of MAGE-A expression as a predictive diagnostic test? Is immunohistochemical or molecular biological (RT-PCR) detection of MAGE-A better suited as a diagnostic test? iii) Can MAGE-A be used successfully as a diagnostic test in practice? iv) Is there an association between MAGE-A expression and immunological changes preceding malignant transformation (macrophage polarization, T cell infiltration, checkpoint expression, TLR expression)? v) Are the immunological changes in OLP potentially amenable to immunomodulatory therapy?

Short summary of the study protocol:

After the patient has been informed and included in the study, the first step is the photo documentation and then the incision biopsy of the OLP. The treating physician is free to choose whether to take a sample from one or more sites of the lesion. This procedure complies with the standard diagnostic guidelines and is not a study-specific measure. Thus, there is no deviation from the clinical routine for the study and no invasive measure required by the study. The sample taken is then divided. The total amount of tissue taken corresponds to the amount taken in the routine outside the study. One part of the sample is conventionally fixed in formalin. The second part (max. 5x5x2mm) is preserved in RNA later for later PCR analysis. Both samples will be sent to the study center in Erlangen. There the histological evaluation of the tissue takes place in the Pathological Institute of the University Hospital Erlangen within routine diagnostics. The result is communicated to the treating physician and the study centre. The immunohistochemical and molecular biological analyses are carried out in the laboratories of the Oral and Maxillofacial Surgery Erlangen. The results of the analyses are not communicated to the attending physician (blinding). A therapy decision is only made on the basis of clinical and classical histological parameters (degree of dysplasia). D0 and D1 lesions are monitored. D2 and D3 lesions are treated surgically or with laser coagulation depending on the decision of the treating physician and patient. This corresponds to the current clinical standard. If the patient rejects the treatment of the lesion and wishes to continue observing its progress, he remains included in the study. The follow-up time during the study period is 3 years (evaluations also after 2 years). After completion of the study a further follow-up of 2 years is planned in order to achieve a total follow-up of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults, consenting male or female patients
* Age 18 - 80 years
* Diagnosis of one or more leukoplakia of the oral cavity

including

* leukoplakia associated wit lichen planus OR
* leukoplakia associated with diseases of the immune system or immunosuppression OR
* leukoplakia associated with a malignoma of other sites (except oral cavity) in the anamnesis
* Existing consent to participation in the study after clarification has been given

Exclusion Criteria:

* clinical evidence of invasive carcinoma of the oral cavity OR
* carcinoma of the oral cavity in the anamnesis OR
* patients unable to give informed consent OR
* rejection of the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically proven leukoplakia (OLP) of the oral cavity (whitish, non-wipeable oral mucosa changes that cannot be attributed to any disease) are to be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dependence of malignant transformation on a MAGE-A based immunoscore | 2 years
  Association of OLP malignant transformation with a MAGE-A based immunoscore. Into this score, the following immunohistochemical and molecular biological parameters determined in biopsies will be integrated:
  * MAGE-A expression
  * Macrophage infiltration and polarization (CD68, CD163)
  * T cell infiltration (CD3, CD8)
  * Altered expression of immune checkpoints and TLR receptors (PD-L1, PD-L2, TLR7) These parameters will be aggregated to an immunoscore
Dependence of malignant transformation on a MAGE-A based immunoscore | 3 years
  Association of OLP malignant transformation with a MAGE-A based immunoscore. Into this score, the following immunohistochemical and molecular biological parameters determined in biopsies will be integrated:
  * MAGE-A expression
  * Macrophage infiltration and polarization (CD68, CD163)
  * T cell infiltration (CD3, CD8)
  * Altered expression of immune checkpoints and TLR receptors (PD-L1, PD-L2, TLR7) These parameters will be aggregated to an immunoscore
Dependence of malignant transformation on a MAGE-A based immunoscore | 5 years
  Association of OLP malignant transformation with a MAGE-A based immunoscore. Into this score, the following immunohistochemical and molecular biological parameters determined in biopsies will be integrated:
  * MAGE-A expression
  * Macrophage infiltration and polarization (CD68, CD163)
  * T cell infiltration (CD3, CD8)
  * Altered expression of immune checkpoints and TLR receptors (PD-L1, PD-L2, TLR7) These parameters will be aggregated to an immunoscore

SECONDARY OUTCOMES:
Frequency of malignant transformation | 2 years
  Frequency of malignant transformation of OLP (determination of the incidence of OSCC in OLP cases)
Frequency of malignant transformation | 3 years
  Frequency of malignant transformation of OLP (determination of the incidence of OSCC in OLP cases)
Frequency of malignant transformation | 5 years
  Frequency of malignant transformation of OLP (determination of the incidence of OSCC in OLP cases)
Dependence of malignant transformation on dysplasia | 2 years
  Dependence of malignant transformation on histologically determined degree of dysplasia (D0-D3)
Dependence of malignant transformation on dysplasia | 3 years
  Dependence of malignant transformation on histologically determined degree of dysplasia (D0-D3)
Dependence of malignant transformation on dysplasia | 5 years
  Dependence of malignant transformation on histologically determined degree of dysplasia (D0-D3)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Weber, MD, DMD, Study Chair — Maxillofacial Surgery Erlangen; Falk Wehrhan, MD, DMD, Study Chair — Maxillofacial Surgery Erlangen; Jutta Ries, PhD, Study Chair — Maxillofacial Surgery Erlangen
Locations (1):
- Universitätsklinikum Erlangen, FAU Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No